CLINICAL TRIAL: NCT05960617
Title: Efficacy and Safety of Empagliflozin in Patients With Glycogen Storage Disease Type Ib
Brief Title: Efficacy and Safety of Empagliflozin in GSD-Ib Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2023-051-2
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Glycogen Storage Disease Type IB
MeSH Terms: conditions — Glycogen Storage Disease IB | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral administration of Empagliflozin (Experimental): All subjects will have a baseline assessment and be prospectively followed up for 12 months to examine their outcome after receiving empagliflozin.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Oral administration of Empagliflozin:
  The starting dose was 0.3 mg/kg/day in 2 divided doses for 3 months. If the subject had an absolute neutrophil count > 1.0 × 10^9/L and clinical improvement (decreased number of infections and/or decreased IBD activity within 3 months), the maintenance dose was maintained.
  If the subject had an absolute neutrophil count < 1.0 × 10^9/L but clinical improvement (decreased number of infections and/or decreased IBD activity within 3 months), the maintenance dose was maintained and reassessed 1 month later.
  If the subject had an absolute neutrophil count < 1.0 × 10^9/L and no clinical improvement (no change in number of infections and/or no change in IBD activity within 3 months), the dose was increased by 0.1 mg/kg/day and reassessed 3 months later.
  Assessments were then performed every 3 months with the same dose modification criteria as above.
  Other Names: Jardiance

SUMMARY:
Empagliflozin Treatment of GSD-1b patients

DETAILED DESCRIPTION:
Glycogen storage disease type Ib (GSD-Ib) is a type of genetic disease with a prevalence of approximately 1 in 500,000. In addition to phenotypes common to GSD-I such as hypoglycemia, hypoglycemia, lactatemia, hyperlipidemia, hyperuricemia, and hepatomegaly, GSD-Ib patients also experience neutropenia and dysfunction, causing infections and inflammatory bowel disease (IBD). At present, the only available treatment for neutropenia in GSD-Ib patients is subcutaneous injection of granulocyte-colony stimulating factor (G-CSF). G-CSF increases the number of neutrophils, but does not improve neutrophil dysfunction, and is also associated with the risk of concurrent splenomegaly and malignancy.

The most recent research findings demonstrated that substantial accumulation of 1,5-anhydroglucitol-phosphate is the cause of neutropenia and neutrophil dysfunction in GSD Ib patients. Empagliflozin, an SGLT2 inhibitor, is an efficient and secure approach of treating neutropenia in these patients by inhibiting renal glucose and 1,5-anhydroglucitol reabsorption. Our study's objective is to assess the efficacy and safety of empagliflozin (Jardiance®) in patients with GSD Ib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with glycogen storage disease type Ib (genetically diagnosed) aged ≥ 1 year and ≤ 50 years;
2. Patients meet the diagnostic criteria for Crohn's disease (CD) based on Expert consensus on the diagnosis and treatment of inflammatory bowel disease in Chinese children (2019) or Consensus opinion on the diagnosis and treatment of inflammatory bowel disease in China (2018), or patients meet the diagnostic criteria for recurrent respiratory tract infection based on Clinical diagnosis and treatment for recurrent respiratory tract infection in Chinese children (2022);
3. Subjects and their guardians/clients (< 18 years old) or subjects (≥ 18 years old) signed the informed consent form.

Exclusion Criteria:

1. Patients with chronic kidney disease (eGFR < 60 ml/min/1.73 m^2) or cirrhosis (Metavir F4);
2. Experiencing symptomatic or severe hypoglycemia within 1 month before the start of this trial;
3. Absolute neutrophil count continued ≥ 1.5 × 10^9/L (≥ 3 tests, each interval ≥ 5 days);
4. Current active urinary tract infection (until urine routine twice negative);
5. Participating other clinical investigators in the past 1 month;
6. Pregnancy, breast-feeding and having a pregnancy plan;
7. Presence of contraindications to empagliflozin therapy (hypersensitivity to empagliflozin, current or history of gangrene, history of recurrent urinary or genital infections);
8. Patients who are not suitable for participating in the clinical investigator or with low compliance in the investigator 's opinion.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Absolute neutrophil count at 1 year | 1 year
  Efficacy of Empaglifozin measured by the change in absolute neutrophil count after 12 months of treatment compared to the period before study
Occurrence of hypoglycemia | 1 year
  Safety and tolerability of Empaglifozin measured by hypoglycemia

SECONDARY OUTCOMES:
Number of infections | 1 year
  Efficacy of Empaglifozin measured by the number of respiratory tract, skin, and urinary tract infections
Inflammatory bowel disease activity | 1 year
  Measured as classical Crohn 's disease activity index (CDAI) for adults (range from 0 to 600; remission <150; mildly active disease 150-219; moderately active disease 220- 450; severely active disease ≥ 450) or pediatric Crohn' s disease activity index (PCDAI) for children (range from 0 to 100; remission <10; mildly active disease 10-27.5; moderately active disease 30-37.5; severely active disease 40-100) after 3, 6, 9, and 12 months of treatment compared to the period before study
Endoscopic scores of inflammatory bowel disease | 1 year
  Measured as difference in Crohn 's Disease Simplified Endoscopic Score (SES-CD) (range from 0 to 17; remission 0-2; mild endoscopic activity 3-6; moderate endoscopic activity 7-15; severe endoscopic activity >15) before and after 1 year of empagliflozin treatment
Change of triglycerides | 1 year
  Measured as change of triglycerides (mmol/L) compared to the period before study
Change of total cholesterol | 1 year
  Measured as change of total cholesterol (mmol/L) compared to the period before study
Change of lactate | 1 year
  Measured as change of lactate (mmol/L) compared to the period before study
Change of uric acid | 1 year
  Measured as change of uric acid (mmol/L) compared to the period before study

CONTACTS AND LOCATIONS:
Overall Officials: Wenjuan Qiu, MD PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No